CLINICAL TRIAL: NCT05212064
Title: High-flow Nasal Cannula Oxygen Therapy and Hypoxia/Desaturation During Percutaneous Radiofrequency Ablation Under Moderate Sedation: A Randomized Clinical Trial
Brief Title: HFNC and Hypoxia/Desaturation During Radiofrequency Ablation Under Moderate Sedation: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiangling, Clinical Resident, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-2022-262
Record Dates: First submitted 2022-01-19; First posted 2022-01-27 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Propofol; Hypoxia; Sedation Complication; Desaturation of Blood
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal cannula group (Sham Comparator): Heated and humidified oxygen of 6 L/minute was supplied via an HFNC
  Interventions: Other: nasal cannula oxygen therapy
- High-flow nasal cannula (HFNC) (Experimental): Heated and humidified oxygen of 40 L/minute was supplied via an HFNC
  Interventions: Device: high-flow oxygen nasal cannula therapy

INTERVENTIONS:
Device: high-flow oxygen nasal cannula therapy — Heated and humidified oxygen of 40L/minute through high-flow nasal cannula (HFNC) therapy machine.
  Arms: High-flow nasal cannula (HFNC)
Other: nasal cannula oxygen therapy — Heated and humidified oxygen of 6L/minute through high-flow nasal cannula (HFNC) therapy machine.
  Arms: Nasal cannula group

SUMMARY:
Background: Propofol based sedated anesthesia was widely used in percutaneous radiofrequency ablation and hypoxia/desaturation is one of the most frequent adverse events during this procedure. No effective methods have been found to prevent hypoxia/desaturation so far. The aim of this study was to evaluate whether the incidence of hypoxia/desaturation was different between the high-flow nasal cannula (HFNC) therapy group (which can provide heated and humidified oxygen up to 60L/minute.) and the nasal cannula group.

Methods: In a randomized, prospective and double-blind study,100 patients undergo percutaneous radiofrequency ablation based on propofol sedation were assigned into two groups: the nasal cannula group (O2 [6 L/minute] was supplied via an HFNC) and the HFNC group (O2 [40 L/minute] was supplied via an HFNC). The primary outcome is the incidence of hypoxia/desaturation during surgery. Other adverse events were also recorded.

DETAILED DESCRIPTION:
After received the approvement of ethics committee of the Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital, approval number IRB-2022-262). The study was registered before patient enrollment in Clinicaltrials.Written informed consent was obtained from all participants. 100 adult patients between 18-75 years, ASA physical state I to III, undergoing percutaneous radiofrequency ablation, were enrolled in this study.

Preoperative arrangements 3-lead electrocardiogram, pulse oximetry and non-invasive blood pressure were measured for basic monitoring. Local anaesthesia was induced by administering 7 ml of 2% lidocaine before the ablation needle was first inserted into the tumour. Then, 0.15 mg/kg oxycodone (diluted to 1 mg/ml with normal saline; Mundipharma, Vantaa, Finland) was administered to both groups. Rescue opioids were administered when the numerical rating scale (NRS) score was greater than 4 or when the patient had obvious, unwanted body movements. The rescue OXY dose was 0.05 mg/kg with the total dose not to exceed 0.25 mg/kg. Blood pressure was measured every 3 minutes as well as 2 minutes after the drug was administered or at the discretion of the anaesthesiologist. All patients remained in the PACU under monitoring for at least 30 minutes until their Aldrete score was between 9 to 10. Mean blood pressure, heart rate, and respiratory rate were recorded. The effect site concentration of propofol is 1.3 ug/ml at the beginning and adjusted at a stepwise of 0.3 ug/ml to maintain a sedation score between 3-4. The depth of sedation was assessed and recorded every 3 minutes by MOAA/S.

ELIGIBILITY:
Inclusion Criteria:

* 18< age < 75 years;
* ASA physical state I and II; .Undergoing percutaneous radiofrequency ablation.

Exclusion Criteria:

* Age < 18 years or older than 75 years;
* America Society of Anesthesiologists (ASA) class >III;
* Allergic to anesthetic solutions;
* Tendency for nose bleeding or coagulation disorders;
* Local infection (eg. mouth, nose, or throat infection);
* Heart disease like congestive heart failure, severe aortic stenosis or mitral stenosis, cardiac surgery involving thoracotomy (eg, coronary artery bypass graft or valve replacement surgery) in the last 6 months; acute myocardial infarction in the last 6 months; acute arrhythmia (including tachycardia and bradycardia) with hemodynamic instability;
* Diagnosed chronic obstructive pulmonary disease (COPD) or other current acute or chronic lung diseases requiring supplemental chronic or intermittent oxygen therapy;
* Increased intracranial pressure;
* Fever, defined as core body temperature >37.5 C;
* Severe anemia (30g/L< hemoglobin <6g/L);
* Emergency surgery;
* Patients refuse to participate;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Hypoxia | Throughout the procedure
  Observe the incidence of hypoxia/desaturation between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, Ph.D, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Wang J, Wu Q, Ding Z, Zhang W, Xie K, Mao X, Fang X. High-flow nasal cannula oxygenation reduces desaturation during percutaneous radiofrequency ablation under moderate sedation. Front Med (Lausanne). 2025 Jul 23;12:1517819. doi: 10.3389/fmed.2025.1517819. eCollection 2025. PMID 40771463